CLINICAL TRIAL: NCT01756313
Title: Optimizing Uptake of Methylaminolevulinat With Fractional Ablative Laser Technique
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Christina Haak, MD, Bispebjerg Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-4-2012-041
Record Dates: First submitted 2012-12-20; First posted 2012-12-25 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Photodynamic Therapy; Ablative Fractional Laser

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser+Methylaminolevulinat (Experimental): It's a single arm. Intervention as described in the detailed description.
  Interventions: Procedure: Laser+Methylaminolevulinat

INTERVENTIONS:
Procedure: Laser+Methylaminolevulinat — It's a single arm study. Intervention as described in detailed description.

SUMMARY:
The objectives of this study is to investigate if pre-treating the skin with an ablative fractional laser that creates small micropores in the skin:

1. Increases the uptake of Methylaminolevulinat (MAL) in the skin.
2. Decreases the required incubation time of MAL when performing photo dynamic therapy.

DETAILED DESCRIPTION:
12 healthy male individuals were included.

On the back, 25 areas measuring 2.8x2.8 cm were marked, plus one control area. We tested 2 variables.

1) Density of laser channels. 2) Methylaminolevulinat (MAL) concentration

1. Laser - Each area was randomized to receiving:

   * no treatment
   * 1% laser channel density
   * 2% laser channel density
   * 5% laser channel density
   * 10% laser channel density
   * 15% laser channel density
2. MAL - Each density was assigned to 4 areas. Within each density category, the four areas were randomized to receive:

   * vehicle
   * 4% MAL
   * 8%MAL
   * 16%MAL

The uptake of MAL was evaluated by fluorescence intensity measured with a florescence camera at t=

* 0min
* 30min
* 1h
* 1.5h 2h 2.5h 3h

ELIGIBILITY:
Inclusion Criteria:

* Male
* >18 years old
* Fitzpatrick skin type I-III
* No UV exposure thee months prior to study
* Signed study consent

Exclusion Criteria:

* Known allergy to substances in MAL or Unguentum M cream.
* Previous keloid
* Use of topical or systemic photosensitizing drug
* Evaluated to not be able to follow treatment protocol

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Fluorescence Intensity | up to 3 hours
  Fluorescence Intensity measured with a fluorescence camera.

OTHER OUTCOMES:
Skin reactions | 24h
  Evaluating skin reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD PhD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Department of Dermatology, Bispebjerg Hospital, Copenhagen, Denmark